CLINICAL TRIAL: NCT03327779
Title: World Bleeding Disorders Registry
Acronym: WBDR
Status: Recruiting | Type: Observational
Sponsor: World Federation of Hemophilia (Other)
Responsible Party: Sponsor
Other Study IDs: WBDR
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hemophilia A; Hemophilia B; Von Willebrand Diseases
MeSH Terms: conditions — Hemophilia A; Hemophilia B; von Willebrand Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The WBDR is an international observational disease registry of patients with hemophilia. It will provide a platform for a network of hemophilia treatment centres (HTCs) around the world to collect uniform and standardized patient data and guide clinical practice. With informed consent from the patient, the WBDR stores anonymous data about the person's disease, such as hemophilia type and severity, symptoms, and treatment.

DETAILED DESCRIPTION:
The WBDR is a prospective, global registry of patients diagnosed with hemophilia A and B. Following the success of a pilot study, implementation of the full scale WBDR is underway. The goals are to enroll at least 200 HTCs from more than 50 countries, and at least 10,000 people with hemophilia, during the first five years, aiming for representation of patients from around the world and from all levels of access to care. Minimal criteria for participation of HTCs include access to reliable internet, human resources for data entry and commitment to long-term enrolment and follow-up of patients. The WBDR database is being developed through a collaboration between the WFH, Karolinska Institute and Health Solutions.

By combining data from countries around the world, the WBDR will provide a large amount of real world data, on which researchers can address important scientific and clinical issues. The World Bleeding Disorders Registry (WBDR) is intended to fill existing gaps in knowledge by collecting real world data on the patient clinical experience around the globe.

ELIGIBILITY:
Inclusion Criteria:

* Patients of participating Hemophilia Treatment Centres with Hemophilia A or B, or von Willebrand Disease

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of participating Hemophilia Treatment Centres with Hemophilia A or B, or von Willebrand Disease.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | 5 years
Number of participating Hemophilia Treatment Centres | 5 years
Number of participating countries | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- World Federation of Hemophilia, Montreal, Quebec, Canada